CLINICAL TRIAL: NCT00167440
Title: Comparison of Techniques for Assessing Cardiac Output and Preload in Critically Ill Patients
Brief Title: Comparison of Techniques for Assessing Cardiac Output and Preload in Critically Ill Pediatric Patients
Status: Withdrawn | Type: Observational
Why Stopped: Personelle changes mandated suspension.
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, jeffrey rubenstein, Professor, University of Rochester
Other Study IDs: 10398; 5R44HL06199403
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Low Cardiac Output
Keywords: cardiac index; cardiac output; indwelling central venous catheter; indwelling arterial catheter
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Each year in the United States more than 30,000 children are admitted to intensive care units. The majority of these children have some degree of heart instability during their stay, yet there is currently no routine way to measure the actual amount of blood that the heart pumps. The ability to measure the amount of blood that the heart pumps accurately and easily at frequent intervals would be very helpful to the doctor caring for these children because many of them have poor heart function as a result of their illnesses. Current techniques used in adults to measure output of the heart are either not readily transferred to children or demand difficult invasive procedures. Because of this, the amount of blood that the heart pumps cannot be measured with enough frequency to help guide care. Despite this reality, accurate measurements of the amount of blood that the heart pumps in these patients at crucial points in their illnesses would allow for more accurate use of potentially harmful procedures and could possibly improve the outlook for these children. Likewise, being able to correctly measure blood volume could provide a better way to estimate the pressure on the heart and improve treatment.

The purpose of this research study is to compare the accuracy of doctor estimates of heart output, and establish the usefulness of central blood volume measurements by PCOM (pediatric cardiac output measurements), a less invasive procedure

DETAILED DESCRIPTION:
The ability to measure cardiac output accurately and reproducibly at frequent intervals remains elusive to the clinician caring for critically ill pediatric patients although a large proportion of these children are known to have hemodynamic compromise as a result of their illnesses. I propose to define the accuracy of clinician estimates of cardiac output in these patients and to test the ability of a new device that measures central blood volume to predict preload in this setting.

I will study 100 patients in two groups. The first group will consist of critically ill pediatric patients at the time of admission to the PICU. These 50 patients will have cardiac output estimated by three methods: Estimation by a "panel of experienced clinicians"; Calculation of the arteriovenous content difference; and Direct measurement using a new minimally invasive system based on assessing changes in ultrasound transmission in blood after intravenous administration of a small (< 5 ml) bolus of normal saline. Group two will consist of 50 PICU patients who therapeutically require either a fluid bolus (25 patients) or a single intravenous dose of diuretic (25 patients). These patients will be assessed in the same fashion at the outset, but will have ongoing measurements of cardiac output and central blood volume using the minimally invasive system and central venous pressure using conventional techniques at 3 intervals within the first hour.

Data will be analyzed to evaluate the strength of correlations between expert assessment and objective measures of cardiac output in all patients (linear regression with calculation of correlation coefficient). Group two patients will be divided according to therapeutic intervention. The strength of correlation between changes in central blood volume and changes in central venous pressure and cardiac output will be assessed using similar statistical techniques.

ELIGIBILITY:
Inclusion Criteria:

* patients less than 16 years of age
* admitted to the PICU after surgery
* indwelling central venous and arterial catheters
* arterial oxygen saturation greater than 94% while breathing 60% oxygen
* ability to draw blood from both arterial and venous catheters
* require fluid bolus or dose of diuretic
* require mechanical ventilation
* no change in dosing of inotropic or vasoactive agents over prior to 60 minutes

Exclusion Criteria:

* hemodynamic instability

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, newborn through age 16 admitted to a pediatric intensive care unit (PICU)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rubenstein, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States